CLINICAL TRIAL: NCT03277144
Title: Does the Technique of Duodenal Resection Affect the Incidence of Duodenal Stump Fistula After Gastrectomy for Gastric Cancer ? A Randomized Controlled Trial (DRTST: Duodenal Resection Tri-staple Technology)
Brief Title: Incidence of Duodenal Stump Fistula After Gastrectomy for Gastric Cancer. A Randomized Controlled Trial
Acronym: DRTST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Maurizio Degiuli, Associate Professor, Head Surgical Oncology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DRTST.01
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer; Duodenal Stump Leak
Keywords: linear stapler
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: All gastric cancer patients who meet the inclusion/exclusion criteria and give the informed consent to participate are registered into the central trial database and centrally permuted-block randomized to one of the two arms (a. Duodenal Stump Closure with TriStaple Technology - TST or b. Duodenal Stump closure with other conventional techniques - OCT ).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TST-TriStaple(3lines stapler)Technology (Experimental): During gastrectomy for gatric cancer without anastomosis with the duodenum, Duodenal Stump is closed with a TriStaple (three-lines linear stapler) Technology device.
  Interventions: Device: TST-TriStaple(3lines stapler)Technology
- OCT (other conventional techniques) (Active Comparator): During gastrectomy for gatric cancer without anastomosis with the duodenum, Duodenal Stump is closed with conventional techniques including manual sutures and devices with only two lines of staples.
  Interventions: Other: other conventional techniques

INTERVENTIONS:
Device: TST-TriStaple(3lines stapler)Technology — Duodenal stump closed using a Tristaple ( three-lines linear stapler) device
  Arms: TST-TriStaple(3lines stapler)Technology
Other: other conventional techniques — Duodenal stump closed using other conventional techniques entailing manual suture or mechanical devices with only two lines of sutures.
  Other Names: double-line linear stapler with manual reinforcement; manual suture; purse string suture; double-line linear stapler without manual reinforcement
  Arms: OCT (other conventional techniques)

SUMMARY:
The goal of this trial is to demonstrate that the use of Tri-Staple Technology for duodenal resection during open gastrectomy for cancer is safer than the use of other conventional methods of resection/closure of the duodenum and that the incidence of duodenal fistula can be decreased to that observed after the use of this technology in Laparoscopic and robotic gastrectomy, therefore almost three times lower than that currently reported in literature.

Participating centres must have an annual volume of at least 20 gastrectomies per year.

DETAILED DESCRIPTION:
BACKGROUND Gastric cancer is still one of the most frequent malignancies in Europe. In United States the estimated new cases in 2010 were 21000 (12730 male and 8270 female) with 10570 estimated deaths (6350 male and 4220 female)[7,8]. In Italy the estimated new cases in 2013 were 13200 (7900 males and 5300 female) (AIOM-AIRTUM, I numeri del cancro in Italia - 2013, www.registri-tumori.it) .The incidence rates in 2005-2009 were 21.6 and 10.8 per 100,000 in males and females respectively. The mortality rates in 2005-2009 were 14.9 and 7.3 per 100,000 in males and females respectively. (www.itacan.ispo.toscana.it).A total or subtotal gastrectomy with D2 lymph node dissection and R0 margins remains the standard of care for gastric cancer[9,10]. Despite this, in low-volume centers gastrectomy still remains a challenging procedure with a notable morbidity rate (33%-43%) and mortality rate (7%-12%)[11,12]. Duodenal stump fistula (DSF) represents an infrequent but severe complication after total or subtotal gastrectomy for gastric cancer, with incidence of 2,5 - 5% and mortality rate ranging from 7% to 67%(1-5). Several factors were identified as possible cause of DSF, such as local hematoma, inflammation, intra-operative inadequate closure of the duodenal stump, incorrect drain position, devascularization, post-operative distension of the duodenum and R1-R2 resections[2,13].

There are many DSF-related complications leading to longer hospitalization times, such as intra-abdominal abscesses, wound infections, diffuse peritonitis, sepsis, malnutrition, pancreatitis, abdominal bleeding, and pneumonia. (3) DSF is often difficult to treat because of the highly enzyme-rich duodenal juice and deep location of the fistula. In a retrospective multicenter study (2) 3,685 patients undergoing gastrectomy for malignancies who developed 68 DSFs were analyzed; it was reported that DSF features had changed in the last 30 years and that DSF alone no longer leads to death; some complications observed in the past, such as fluid and electrolyte loss and dermatitis, have disappeared owing to improvements( in particular parenteral nutrition and wound care). However, additional new complications such as bleeding and fistulas of neighboring organs were emerging. Although medical therapy is associated with better outcomes, surgery is still mandatory in cases of severe abdominal sepsis or bleeding not otherwise manageable.

However, reoperation is often ineffective owing to postoperative edema and inflammation, and the prognosis of patients undergoing surgery for DSF remains very poor. To improve the outcome of these patients, many surgical procedures have been proposed from washing the peritoneal cavity and abdominal drainage to tube duodenostomy (14,15), closure of the fistula, fistula repair with a rectus abdominis flap (16), fistula closure by Roux-en-Y duodenojejunostomy(17,18), biliogastric diversion, laparostomy, and pancreatoduodenectomy (19) but surgeons are often unsure about the best management and the result are often unsuccessful.

In a recent Korean national RCT (6) on open (ODG) vs laparoscopic distal gastrectomy (LADG), the incidence of duodenal stump leakage after laparoscopyc gastrectomy was about 1%; in this population study the use of tri-staple technology for duodenal resection was mandatory. In our clinical practice, the incidence of DSF after open gastrectomy is about 3-5% adopting different techniques of duodenal stump resection/closure.

The aim of this study is to evaluate if duodenal stump resection/closure using tri-staple technology can significantly decrease the incidence of DSF after open gastrectomy as compared to the other conventional methods adopted in the clinical practice (1% vs 5%).

We have designed a national multicentre pragmatic (20) RCT to compare the use of endoGIA or Echelon (triStaple technology) to other conventional methods (GIA with or without manual reinforcement , manual suture, purse string) for duodenal resection/closure during open gastrectomy, with the assumption that Tri-staple technology without reinforcement ( as routinely used in LADG) is the safest method.

AIM OF THE STUDY The goal of this trial is to demonstrate that the use of Tri-Staple Technology for duodenal resection during open gastrectomy for cancer is safer than the use of other conventional methods of resection/closure of the duodenum and that the incidence of duodenal fistula can be decreased to that observed after the use of this technology in Laparoscopic and robotic gastrectomy, therefore almost three times lower than that currently reported in literature.

Participating centres must have an annual volume of at least 20 gastrectomies per year.

Design of the study This is a multicentre randomized controlled trial.

Patients with malignant tumor of the stomach, as primary diagnosis, requiring distal or total gastrectomy without anastomosis with the duodenum will undergo clinical preoperative workout and anaesthesiologist evaluation. All patients who meet the inclusion/exclusion criteria and agree to sign the informed consent are registered into the trial and randomized to one of the two arms (a. Duodenal Stump Closure with TriStaple Technology - TST or b. Duodenal Stump closure with other conventional techniques - OCT ) as described in the chapter Randomization. In TST arm no manual reinforce of the mechanical suture should be perfomed; in OCT group, a manual reinforce of the suture can be done according to the preference of the operator, and recorded in the trial data base (DB).

Patients' postoperative course will be carefully monitored and all variables detailed below will be recorded in the DB.

DSF will be diagnosed by the presence of duodenal fluid in the surgical drainage and confirmed by a CT scan when needed (presence of intra-abdominal peri-duodenal collection of fluid and/or micro air bubbles).

Also the type of treatment (conservative, percutaneous drainage, reoperation, others ) of DSF should be recorded, as well as the length of hospital stay and other postoperative complications or in-hospital death ( as well as 30- and 90- days mortality)

Trial setting

This is an Italian national multicentre RCT; the Division of General Surgery from University of Turin, Department of Surgical Sciences, AOU San Luigi Gonzaga di Orbassano, will be the Coordinating Centre of the trial. The P.I. of the trial is Prof Maurizio Degiuli.

S.S.D. Epidemiologia, Clinica e Valutativa, AOU Città della Salute e della Scienza di Torino, will be responsible for this trial's central randomisation and statistical analysis.

Clinical monitoring and data managing will be performed by the P.I. and and co-investigators.

Study population

inclusion criteria

pathologically proven malign tumor of the stomach age of 18 to 80 years, no history of other cancers no history of radiotherapy in supra-mesocolic space total or distal gastrectomy without anastomosis with the duodenum

exclusion criteria

emergency surgery American Society of Anesthesiologists class > 3 need for combined resection of other organs laparoscopic/robotic access severe heart disease liver cirrhosis T stage >cT4a citology positive at preoperative laparoscopy cM+ cD+

All patients freely give informed consent to participate in the study prior to surgery, at the time of discussing the intervention with the surgeon or the nurse and can decide to withdraw from the study at any time.

Diagnosis of DSF

A diagnosis of DF is made on the basis of the presence of duodenal juice in the surgical drainage or its leakage through the abdominal wall, and confirmed by CT scan and/or fistulography.

Variables

sex age ASA score COPD type 2 DM multiple comorbidities pre-operative albumin serum levels pre-operative lymphocytes blood count cT Stage / pTStage pTNM distal margin involvement intraoperative blood loss lenght of hospital stay Type of gastrectomy TG vs DG type of reconstruction: ( BII vs RY) lymph node dissection: D1, D1+, D2, > D2

Type of duodenal stump closure device:

A. endoGIA tristaple B. other techniques (GIA/TA with or without manual reinforcement (simple interrupted suture or running suture), manual suture (simple interrupted or running suture), purse string)

Development of DSF (po day) healing of DSF (po day) Diagnosis of DSF Daily output of DSF Type of treatment of DSF Other postoperative morbidity according to Dindo. Postoperative mortality

Randomisation

All patients who meet the inclusion/exclusion criteria and give the informed consent to participate are registered into the central trial database and centrally randomized to one of the two groups (a. Duodenal Stump Closure with TriStaple Technology - TST or b. Duodenal Stump closure with other conventional techniques - OCT ).

Patients refusing recruitment are treated with usual care and contribute to the database a limited set of pre-defined information.

Result of randomisation is communicated to the surgical team at the time of their entrance in the surgical theatre.

Sample size calculation and statistical analysis

Assuming an alpha error at the 5% level and power 80%, a total of 700 patients (350 per arm) are required in order to recognise a true difference of 5% in (a) vs 1% in (b).

Assuming an average case volume of 20 patients per year and 60% acceptance rate, about 30 Centres recruiting for two years will need to be involved.

Cox regression with multivariable analysis will be performed

Data property

Results will be the property of Università degli studi di Torino and of the researchers involved in the conduction of the mulicentre project. A scientific committee will be constituted comprising a lead investigator from each of the Centres.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven malign tumor of the stomach
* age of 18 to 80 years,
* no history of other cancers
* no history of radiotherapy in supra-mesocolic space
* total or distal gastrectomy without anastomosis with the duodenum

Exclusion Criteria:

* emergency surgery
* American Society of Anesthesiologists class > 3
* need for combined resection of other organs
* laparoscopic/robotic access
* severe heart disease
* liver cirrhosis
* T stage >cT4a
* citology positive at preoperative laparoscopy
* cM+ (clinical suspicion of distant metastasis)
* cD+ (clinical suspicion of duodenal involvment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-09-11 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
incidence of duodenal stump leak | within 30/60 days from operation
  The aim of this study is to evaluate if duodenal stump closure using tri-staple technology can significantly decrease the incidence of duodenal stump leakage to 1% as compared to other conventional methods (5%). So the primary endpoint is :
  - incidence of DSF, diagnosed on the basis of the presence of duodenal juice in the surgical drainage or its leakage through the abdominal wall, and confirmed by CT scan and/or fistulography.

SECONDARY OUTCOMES:
cost of surgery | within 90 days from operation
  cost of devices, hospital stay, drugs, examinations
operative time for duodenal stump closure | intraopeartively
  time ( min) necessary for duodenal stump closure
short-term postoperative complications | within 30 days from operation
  onset of postoperative complications according to Clavien-Dindo classification
blood loss | intraopeartively
  intraoperative blood loss (ml)
lenght of hospitalization | 120 days after operation
  duration (days) of hospital stay after operation
Operative mortality | 30 and 60 days after operation
  post-operative death
Frequency of DSF by surgical volume | one year
  rate of duodenal stump leak of every participating center

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Degiuli, MD Prof, Principal Investigator — University of Turin, San Luigi University Hospital
Locations (1):
- San Luigi University Hospital, Orbassano, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inghelmann R, Grande E, Francisci S, Verdecchia A, Micheli A, Baili P, Capocaccia R, De Angelis R. Regional estimates of stomach cancer burden in Italy. Tumori. 2007 Jul-Aug;93(4):367-73. doi: 10.1177/030089160709300407. PMID 17899867
- [Background] Aurello P, Bellagamba R, Rossi Del Monte S, D'Angelo F, Nigri G, Cicchini C, Ravaioli M, Ramacciato G. Apoptosis and microvessel density in gastric cancer: correlation with tumor stage and prognosis. Am Surg. 2009 Dec;75(12):1183-8. PMID 19999909
- [Background] Aurello P, Magistri P, Nigri G, Petrucciani N, Novi L, Antolino L, D'Angelo F, Ramacciato G. Surgical management of microscopic positive resection margin after gastrectomy for gastric cancer: a systematic review of gastric R1 management. Anticancer Res. 2014 Nov;34(11):6283-8. PMID 25368226
- [Background] Martin RC 2nd, Jaques DP, Brennan MF, Karpeh M. Achieving RO resection for locally advanced gastric cancer: is it worth the risk of multiorgan resection? J Am Coll Surg. 2002 May;194(5):568-77. doi: 10.1016/s1072-7515(02)01116-x. PMID 12025834
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Result] Orsenigo E, Bissolati M, Socci C, Chiari D, Muffatti F, Nifosi J, Staudacher C. Duodenal stump fistula after gastric surgery for malignancies: a retrospective analysis of risk factors in a single centre experience. Gastric Cancer. 2014 Oct;17(4):733-44. doi: 10.1007/s10120-013-0327-x. Epub 2014 Jan 8. PMID 24399492
- [Result] Cozzaglio L, Coladonato M, Biffi R, Coniglio A, Corso V, Dionigi P, Gianotti L, Mazzaferro V, Morgagni P, Rosa F, Rosati R, Roviello F, Doci R. Duodenal fistula after elective gastrectomy for malignant disease : an italian retrospective multicenter study. J Gastrointest Surg. 2010 May;14(5):805-11. doi: 10.1007/s11605-010-1166-2. Epub 2010 Feb 9. PMID 20143272
- [Result] Rossi JA, Sollenberger LL, Rege RV, Glenn J, Joehl RJ. External duodenal fistula. Causes, complications, and treatment. Arch Surg. 1986 Aug;121(8):908-12. doi: 10.1001/archsurg.1986.01400080050009. PMID 3729708
- [Result] EDMUNDS LH Jr, WILLIAMS GM, WELCH CE. External fistulas arising from the gastro-intestinal tract. Ann Surg. 1960 Sep;152(3):445-71. doi: 10.1097/00000658-196009000-00009. No abstract available. PMID 13725742
- [Result] Tarazi R, Coutsoftides T, Steiger E, Fazio VW. Gastric and duodenal cutaneous fistulas. World J Surg. 1983 Jul;7(4):463-73. doi: 10.1007/BF01655935. No abstract available. PMID 6624121
- [Result] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Result] Pedrazzani C, Marrelli D, Rampone B, De Stefano A, Corso G, Fotia G, Pinto E, Roviello F. Postoperative complications and functional results after subtotal gastrectomy with Billroth II reconstruction for primary gastric cancer. Dig Dis Sci. 2007 Aug;52(8):1757-63. doi: 10.1007/s10620-006-9655-6. Epub 2007 Apr 3. PMID 17404848
- [Result] McCulloch P, Ward J, Tekkis PP; ASCOT group of surgeons; British Oesophago-Gastric Cancer Group. Mortality and morbidity in gastro-oesophageal cancer surgery: initial results of ASCOT multicentre prospective cohort study. BMJ. 2003 Nov 22;327(7425):1192-7. doi: 10.1136/bmj.327.7425.1192. PMID 14630753
- [Result] Cozzaglio L, Cimino M, Mauri G, Ardito A, Pedicini V, Poretti D, Brambilla G, Sacchi M, Melis A, Doci R. Percutaneous transhepatic biliary drainage and occlusion balloon in the management of duodenal stump fistula. J Gastrointest Surg. 2011 Nov;15(11):1977-81. doi: 10.1007/s11605-011-1668-6. Epub 2011 Sep 13. PMID 21913043
- [Result] Levy E, Cugnenc PH, Frileux P, Hannoun L, Parc R, Huguet C, Loygue J. Postoperative peritonitis due to gastric and duodenal fistulas. Operative management by continuous intraluminal infusion and aspiration: report of 23 cases. Br J Surg. 1984 Jul;71(7):543-6. doi: 10.1002/bjs.1800710725. PMID 6733430
- [Result] Isik B, Yilmaz S, Kirimlioglu V, Sogutlu G, Yilmaz M, Katz D. A life-saving but inadequately discussed procedure: tube duodenostomy. Known and unknown aspects. World J Surg. 2007 Aug;31(8):1616-24; discussion 1625-6. doi: 10.1007/s00268-007-9114-3. PMID 17566821
- [Result] Chander J, Lal P, Ramteke VK. Rectus abdominis muscle flap for high-output duodenal fistula: novel technique. World J Surg. 2004 Feb;28(2):179-82. doi: 10.1007/s00268-003-7017-5. Epub 2004 Jan 20. PMID 14727065
- [Result] Ujiki GT, Shields TW. Roux-en-Y operation in the management of postoperative fistula. Arch Surg. 1981 May;116(5):614-7. doi: 10.1001/archsurg.1981.01380170094017. PMID 7235954
- [Result] Milias K, Deligiannidis N, Papavramidis TS, Ioannidis K, Xiros N, Papavramidis S. Biliogastric diversion for the management of high-output duodenal fistula: report of two cases and literature review. J Gastrointest Surg. 2009 Feb;13(2):299-303. doi: 10.1007/s11605-008-0677-6. Epub 2008 Sep 30. PMID 18825468
- [Result] Musicant ME, Thompson JC. The emergency management of lateral duodenal fistula by pancreaticoduodenectomy. Surg Gynecol Obstet. 1969 Jan;128(1):108-14. No abstract available. PMID 5774989